CLINICAL TRIAL: NCT01750190
Title: A Phase 3, Randomized, Double-Blind, Placebo Controlled Study of the Efficacy and Safety of Roxadustat (FG-4592) for the Treatment of Anemia in Chronic Kidney Disease Patients Not on Dialysis
Brief Title: A Study of Roxadustat for the Treatment of Anemia in Participants With Chronic Kidney Disease and Not Receiving Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-4592-060
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: CKD Anemia
Keywords: anemia; chronic kidney disease (CKD); non-dialysis; Hemoglobin (Hb); End-Stage Renal Disease; erythropoeitin; ASP1517; erythropoeisis stimulating-agent; AZD9941
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental): Participants will receive roxadustat tablets orally 3 times a week (TIW). The initial dose will be according to the tiered weight-based approach, with starting roxadustat doses of 70 milligrams (mg) TIW to participants weighing <70 kilograms (kg) and roxadustat doses of 100 mg TIW to participants weighing ≥70 kg. Dose-titration (up to a maximum dose of 300 mg) will be performed based upon regular measurement of Hb levels until the participant achieves central Hb value of ≥11.0 grams/deciliter (g/dL) and Hb increase from baseline (BL) of ≥1.0 g/dL at 2 consecutive study visits, separated by at least 5 days. Once target Hb level is reached, the participant will enter the maintenance period during which roxadustat dosage will be adjusted every 4 weeks to maintain participant's Hb level within the target range of 10.0 g/dL and 12.0 g/dL. The maximum treatment duration will be up to 234.9 weeks.
  Interventions: Drug: Roxadustat
- Placebo (Placebo Comparator): Participants will receive roxadustat-matching placebo tablets orally TIW. The initial dose will be according to the tiered weight-based approach, with starting roxadustat-matching placebo doses of 70 mg TIW to participants weighing <70 kg and roxadustat-matching placebo doses of 100 mg TIW to participants weighing ≥70 kg. Dose-titration (up to a maximum dose of 300 mg) will be performed based upon regular measurement of Hb levels until the participant achieves central Hb value of ≥11.0 g/dL and Hb increase from BL of ≥1.0 g/dL at 2 consecutive study visits, separated by at least 5 days. Once target Hb level is reached, the participant will enter the maintenance period during which roxadustat dosage will be adjusted every 4 weeks to maintain participant's Hb level within the target range of 10.0 g/dL and 12.0 g/dL. The maximum treatment duration will be up to 208.1 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roxadustat — Oral tablets
  Other Names: FG-4592; ASP1517; AZD9941
  Arms: Roxadustat
Drug: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether roxadustat is safe and effective in the treatment of anemia in participants with chronic kidney disease and not on dialysis.

DETAILED DESCRIPTION:
There is a screening period of up to 6 weeks, a variable treatment period for individual participants. In order to complete the treatment period simultaneously for all study participants, the minimum treatment duration may be less than 52 weeks, with a maximum treatment duration of up to 3 years after the last participant is randomized, and a post-treatment follow-up period of 4 weeks. Participants who prematurely discontinued from treatment will be expected to complete the Early Termination (ET) and End of Study (EOS) visits. Such participants will be considered non-completers, but they will be expected to participate in long-term follow-up (LTFU) for cardiovascular events (CV) of interest, vital status, and hospitalizations until overall study closure unless the participant withdrew consent for this LTFU data collection. Participants were randomized in a 2:1 ratio to receive either roxadustat or placebo in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease Stages 3, 4, or 5 and not receiving dialysis
* Anemia qualified by measurements of hemoglobin values during screening
* Additional blood work must be in a safe range for study entry
* Body weight 45 to 160 kilograms (kg)
* Willingness to use contraception if of child-bearing potential

Exclusion Criteria:

* Treatment with an erythropoiesis-stimulating agent (ESA) within 12 weeks prior to study participation
* More than 1 dose of intravenous iron within 12 weeks prior to study participation
* Blood transfusion within 8 weeks prior to study participation
* Active infection
* Chronic liver disease
* Severe congestive heart failure, recent heart attack, stroke, seizure, or blood clot
* Uncontrolled blood pressure within 2 weeks prior to study participation
* Renal cell carcinoma
* History of malignancy, including multiple myeloma or other myelodysplastic syndrome
* Chronic inflammatory disease that could impact red blood cell production
* Any prior organ transplant or a scheduled organ transplantation
* Anticipated elective surgery that is expected to lead to significant blood loss or anticipated elective heart procedure
* Gastrointestinal bleeding
* Any prior treatment with roxadustat or a hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI)
* Recent use of an investigational drug or treatment, or participation in an investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 922 (Actual)
Dates: Start 2012-11-05 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Eisner, MD, MPH, Study Chair — Kyntra Bio
Locations (121):
- United States (51):
  - Investigational Site, Huntsville, Alabama
  - Investigational Site, Tempe, Arizona
  - Investigational Site, Alhambra, California
  - Investigational Site, Chula Vista, California
  - Investigational Site, Inglewood, California
  - Investigational Site, La Mesa, California
  - Investigational Site, La Palma, California
  - Investigational Site, Lynwood, California
  - Investigational Site, Northridge, California
  - Investigational Site, Paramount, California
  - Investigational Site, Riverside, California
  - Investigational Site, Roseville, California
  - Investigational Site, San Dimas, California
  - Investigational Site, Whittier, California
  - Investigational Site, Coral Gables, Florida
  - Investigational Site, Cutler Bay, Florida
  - Investigational Site, Hialeah, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, Ocala, Florida
  - Investigational Site, Pembroke Pines, Florida
  - Investigational Site, South Miami, Florida
  - Investigational Site, Winter Park, Florida
  - Investigational Site, Augusta, Georgia
  - Investigational Site, Caldwell, Idaho
  - Investigational Site, Shreveport, Louisiana
  - Investigational Site, Baltimore, Maryland
  - Investigational Site, Boston, Massachusetts
  - Investigational Site, Detroit, Michigan
  - Investigational Site, Flint, Michigan
  - Investigational Site, Pontiac, Michigan
  - Investigational Site, Roseville, Michigan
  - Investigational Site, St Louis, Missouri
  - Investigational Site, New Brunswick, New Jersey
  - Investigational Site, Albuquerque, New Mexico
  - Investigational Site, Mineola, New York
  - Investigational Site, The Bronx, New York
  - Investigational Site, Asheville, North Carolina
  - Investigational Site, Raleigh, North Carolina
  - Investigational Site, Rocky Mount, North Carolina
  - Investigational Site, Winston-Salem, North Carolina
  - Investigational Site, Beaver, Pennsylvania
  - Investigational Site, Orangeburg, South Carolina
  - Investigational Site, Sumter, South Carolina
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Arlington, Texas
  - Investigational Site, Corsicana, Texas
  - Investigational Site, Dallas, Texas
  - Investigational Site, Houston, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site, Fairfax, Virginia
  - Investigational Site, Morgantown, West Virginia
- Argentina (14):
  - Investigational Site, Ciudad Evita, Buenos Aires
  - Investigational Site, González Catán, Buenos Aires
  - Investigational Site, Junín, Buenos Aires
  - Investigational Site, Morón, Buenos Aires
  - Investigational Site, Pergamino, Buenos Aires
  - Investigational Product, Villa Domínico, Buenos Aires
  - Investigational Site, Córdoba, Córdoba Province
  - Investigational Site, Buenos Aires
  - Investigational Site, Corrientes
  - Investigational Site, Córdoba
  - Investigational site, Córdoba
  - Investigational Site, Mendoza
  - Investigational Site, Salta
  - Investigational Site, Santa Fe
- Australia (7):
  - Investigational Site, Liverpool, New South Wales
  - Investigational Site, Gosford
  - Investigational Site, Hobart
  - Investigational Site, Launceston
  - Investigational Site, Melbourne
  - Investigational Site, New Lambton Heights
  - Investigational Site, Randwick
- Chile (2):
  - Investigational Site, Temuco, Región de la Araucanía
  - Investigational Site, Santiago, Santiago Metropolitan
- Colombia (2):
  - Investigational Site, Barranquilla, Atlántico
  - Investigational Site, Bogota, Cundinamarca
- Hong Kong (4):
  - Investigational Site, Hong Kong, Pokfulam
  - Investigational Site, Chai Wan
  - Investigational Site, Shatin
  - Investigational Site, Tai Po
- Malaysia (7):
  - Investigational Site, Alor Star
  - Investigational Site, Kajang
  - Investigational Site, Kuala Lumpur
  - Investigational Site, Kuching
  - Investigational Site, Pulau Pinang
  - Investigational Site, Sungai Petani
  - Investigational Site, Taiping
- Mexico (6):
  - Investigational Site, Guadalajara, Jalisco
  - Investigational Site, Mexico City, Mexico City
  - Investigational Site, Monterrey, Nuevo León
  - Investigational Site, Mérida, Yucatán
  - Investigational Site, Aguascalientes
  - Investigational Site, San Luis Potosí City
- New Zealand (3):
  - Investigational Site, Auckland
  - Investigational Site, Hamilton
  - Investigational Site, Tauranga
- Peru (4):
  - Investigational Site, San Martín de Porres, Lima region
  - Investigational Site, Bellavista, Provincia Constitucional del Callao
  - Investigational site, Lima
  - Investigational Site, Lima
- Philippines (4):
  - Investigational Site, Dasmariñas, Cavite
  - Investigational Site, Davao City, Davao Region
  - Investigational site, Pasig
  - Investigational Site, Quezon City
- Puerto Rico (2):
  - Investigational Site, Ponce
  - Investigational Site, San Juan
- Investigational Site, Singapore, Singapore
- South Korea (6):
  - Investigational Site, Anyang-si, Gyeonggi-do
  - Investigational Site, Goyang-si, Gyeonggi-do
  - Investigational Site, Guri-si, Gyeonggi-do
  - Investigational Site, Seongnam-si, Gyeonggi-do
  - Investigational Site, Busan
  - Investigational Site, Seoul
- Taiwan (6):
  - Investigational Site, Changhua
  - Investigational Site, Hualien City
  - Investigational Site, Kaohsiung City
  - Investigational Site, Taichung
  - Investigational Site, Tainan
  - Investigational Site, Taipei
- Thailand (2):
  - Investigational Site, Bangkok
  - Investigational Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Provenzano R, Szczech L, Leong R, Saikali KG, Zhong M, Lee TT, Little DJ, Houser MT, Frison L, Houghton J, Neff TB. Efficacy and Cardiovascular Safety of Roxadustat for Treatment of Anemia in Patients with Non-Dialysis-Dependent CKD: Pooled Results of Three Randomized Clinical Trials. Clin J Am Soc Nephrol. 2021 Aug;16(8):1190-1200. doi: 10.2215/CJN.16191020. PMID 34362786
- [Derived] Coyne DW, Roger SD, Shin SK, Kim SG, Cadena AA, Moustafa MA, Chan TM, Besarab A, Chou W, Bradley C, Eyassu M, Leong R, Lee TT, Saikali KG, Szczech L, Yu KP. Roxadustat for CKD-related Anemia in Non-dialysis Patients. Kidney Int Rep. 2020 Dec 5;6(3):624-635. doi: 10.1016/j.ekir.2020.11.034. eCollection 2021 Mar. PMID 33732977

RESULTS

PARTICIPANT FLOW:
Groups:
- Roxadustat: Participants received roxadustat tablets orally 3 times a week (TIW). The initial dose was according to the tiered weight-based approach, with starting roxadustat doses of 70 milligrams (mg) TIW to participants weighing <70 kilograms (kg) and roxadustat doses of 100 mg TIW to participants weighing ≥70 kg. Dose-titration (up to a maximum dose of 300 mg) was performed based upon regular measurement of Hb levels until the participant achieved central Hb value of ≥11.0 grams/deciliter (g/dL) and Hb increase from baseline (BL) of ≥1.0 g/dL at 2 consecutive study visits, separated by at least 5 days. Once target Hb level was reached, the participant entered the maintenance period during which roxadustat dosage will be adjusted every 4 weeks to maintain participant's Hb level within the target range of 10.0 g/dL and 12.0 g/dL. The maximum treatment duration was 234.9 weeks.
- Placebo: Participants received roxadustat-matching placebo tablets orally TIW. The initial dose was according to the tiered weight-based approach, with starting roxadustat-matching placebo doses of 70 mg TIW to participants weighing <70 kg and roxadustat-matching placebo doses of 100 mg TIW to participants weighing ≥70 kg. Dose-titration (up to a maximum dose of 300 mg) was performed based upon regular measurement of Hb levels until the participant achieved central Hb value of ≥11.0 g/dL and Hb increase from BL of ≥1.0 g/dL at 2 consecutive study visits, separated by at least 5 days. Once target Hb level was reached, the participant entered the maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participant's Hb level within the target range of 10.0 g/dL and 12.0 g/dL. The maximum treatment duration was 208.1 weeks.
Period: Overall Study
Arm/Group | Roxadustat | Placebo
Started (Intent-to-Treat (ITT) Population: All randomized/enrolled participants.) | 616 | 306
Safety Population (All randomized/enrolled participants who received at least 1 dose of study drug.) | 611 | 305
Full Analysis Set (FAS) (All randomized/enrolled participants who received at least 1 dose of study drug and have baseline and at least 1 postdose Hb assessment.) | 608 | 305
Completed | 349 | 98
Not Completed | 267 | 208
Not completed — Adverse Event | 47 | 19
Not completed — Death | 38 | 11
Not completed — Lack of Efficacy (Including Erythropoiesis-Stimulating Agent Rescue) | 2 | 43
Not completed — Lost to Follow-up | 28 | 7
Not completed — Physician Decision | 16 | 17
Not completed — Protocol Violation | 6 | 5
Not completed — Study/Site Terminated by Sponsor | 4 | 1
Not completed — Withdrawal by Subject | 83 | 89
Not completed — Kidney Transplant | 8 | 4
Not completed — Dialysis | 22 | 8
Not completed — Other than Specified | 13 | 4

BASELINE CHARACTERISTICS:
Population: ITT Population included all randomized/enrolled participants.
Groups:
- Roxadustat: Participants received roxadustat tablets orally TIW. The initial dose was according to the tiered weight-based approach, with starting roxadustat doses of 70 mg TIW to participants weighing <70 kg and roxadustat doses of 100 mg TIW to participants weighing ≥70 kg. Dose-titration (up to a maximum dose of 300 mg) was performed based upon regular measurement of Hb levels until the participant achieved central Hb value of ≥11.0 g/dL and Hb increase from BL of ≥1.0 g/dL at 2 consecutive study visits, separated by at least 5 days. Once target Hb level was reached, the participant entered the maintenance period during which roxadustat dosage will be adjusted every 4 weeks to maintain participant's Hb level within the target range of 10.0 g/dL and 12.0 g/dL. The maximum treatment duration was 234.9 weeks.
- Total: Total of all reporting groups
Arm/Group | Roxadustat | Placebo | Total
Number analyzed (Participants) | 616 | 306 | 922
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 271 | 146 | 417
  >=65 years | 345 | 160 | 505
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 375 | 176 | 551
  Male | 241 | 130 | 371
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 165 | 84 | 249
  Not Hispanic or Latino | 451 | 222 | 673
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/ Alaskan Native | 6 | 1 | 7
  Asian | 310 | 151 | 461
  Black/African American | 76 | 28 | 104
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  White | 176 | 99 | 275
  Other | 46 | 23 | 69

OUTCOME MEASURES:

1. Primary Outcome: United States (US FDA) Submission: Mean Change From Baseline in Hb (g/dL) Over Weeks 28 to 52 Regardless of Rescue Therapy
Description: The change in Hb from baseline to the average level during the evaluation period (defined as Week 28 until Week 52) is reported. Hb values under the influence of a rescue therapy were not censored. The intermittent missing hemoglobin data were imputed for each treatment relying on non-missing data from all participants within each treatment group using the Monte Carlo Markov Chain (MCMC) imputation model, Monotone missing data were imputed by regression from its own treatment group. Baseline Hb was defined as the mean of up to 4 last central laboratory values prior to the first dose of study drug.
Time Frame: Baseline (Day 1, Week 0), Weeks 28 to 52
Population: ITT Population included all randomized/enrolled participants.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 616 | 306
g/dL
  Baseline | 9.10 (0.75) | 9.09 (0.69)
  Change at Weeks 28 to 52 | 2.00 (0.952) | 0.16 (0.895)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Treatment comparison was made using the multiple imputation strategy by combining the results of analysis of covariance (ANCOVA) model with baseline Hb and baseline estimated glomerular filtration rate (eGFR) as covariates and treatment and other randomization stratification factors, except baseline Hb (≤8 g/dL versus >8 g/dL) and eGFR (<30 versus ≥30 milliliters [mL]/minutes [min]/1.73 meters [m]^2), as fixed effects; Test type: Superiority; p < 0.0001, ANCOVA; MI (Multiple Imputation) ANCOVA; Least Square Mean Difference = 1.85, 95% CI 2-sided [1.735 to 1.967], Standard Error of Mean 0.059 — Roxadustat - Placebo Treatment Difference

2. Primary Outcome: Ex-US Submission: Number (%) of Participants Who Achieved a Hb Response During the First 24-Weeks of Treatment Censoring for Rescue Therapy
Description: The number of participants who achieved a Hb response at 2 consecutive visits at least 5 days apart during the first 24 weeks of treatment, without rescue therapy (that is, red blood cell [RBC] transfusion, erythropoiesis-stimulating agent [ESA], or intravenous [IV] iron) are reported. A Hb response is defined, using central laboratory values, as the following:
  * Hb ≥11 g/dL and Hb increase from baseline by ≥1 g/dL in participants with baseline Hb >8 g/dL, or
  * An increase in Hb by ≥2 g/dL in participants with baseline Hb ≤8.0 g/dL
Time Frame: Baseline up to Week 24
Population: FAS Population included of all randomized/enrolled participants who received at least 1 dose of study drug and had baseline and at least 1 postdose Hb assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
Participants | 523 | 20
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 77.56, 95% CI 2-sided [44.73 to 134.48] — Roxadustat/Placebo Odds ratio

3. Secondary Outcome: Mean Change From Baseline in Hb Averaged Over Weeks 28 to 36 With Censoring for Rescue Therapy
Description: For Ex-US submission only: Hb values under the influence of a rescue therapy were censored by mixed effect model of repeated measures (MMRM) for up to 6 weeks. Baseline Hb was defined as the mean of up to 4 last central laboratory values prior to the first dose of study drug.
Time Frame: Baseline (Day 1, Week 0), Weeks 28 to 36
Population: FAS Population included all randomized/enrolled participants who received at least 1 dose of study drug and had baseline and at least 1 postdose Hb assessment. Here, 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
g/dL
  Baseline | 9.09 (0.749) | 9.09 (0.694)
  Change at Weeks 28 to 36: number analyzed (Participants) | 520 | 219
  Change at Weeks 28 to 36 | 2.02 (1.067) | 0.20 (0.994)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Treatment comparison was made using MMRM with baseline Hb and baseline eGFR as covariates, and treatment, visit, visit-by-treatment interaction, and the randomization stratification factors, except baseline Hb (≤8 g/dL versus >8 g/dL) and eGFR (<30 versus ≥30 mL/min/1.73m^2), as fixed effects; Test type: Superiority; p < 0.0001, Mixed Models Analysis; MMRM Analysis; Least Square Mean Difference = 1.88, 95% CI 2-sided [1.730 to 2.037], Standard Error of Mean 1.88 — Roxadustat - placebo treatment difference

4. Secondary Outcome: Mean Change From Baseline in Hb Averaged Over Weeks 28 to 52 Regardless of Rescue Therapy in Participants With Baseline C-Reactive Protein (CRP) >Upper Limit of Normal (ULN)
Description: Hb values under the influence of a rescue therapy were not censored in the analysis. The intermittent missing hemoglobin data were imputed for each treatment relying on non-missing data from all participants within each treatment group using the MCMC imputation model, Monotone missing data were imputed by regression from its own treatment group. Baseline Hb was defined as the mean of up to 4 last central laboratory values prior to the first dose of study treatment.
Time Frame: Baseline (Day 1, Week 0), Weeks 28 to 52
Population: FAS Population included all randomized/enrolled participants who received at least 1 dose of study drug and had baseline and at least 1 postdose Hb assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 156 | 81
g/dL
  Baseline | 9.10 (0.750) | 8.99 (0.668)
  Change at Weeks 28 to 52 | 2.02 (0.933) | 0.18 (0.946)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Treatment comparison was made using the multiple imputation strategy by combining the results of ANCOVA model with baseline Hb and baseline eGFR as covariates , and treatment and other randomization stratification factors, except baseline Hb (≤8 g/dL versus >8 g/dL) and eGFR (<30 versus ≥30 mL/min/1.73m^2 ), as fixed effects; Test type: Superiority; p < 0.0001, ANCOVA; MI ANCOVA; Least Square Mean Difference = 1.90, 95% CI 2-sided [1.663 to 2.143], Standard Error of Mean 0.122 — Roxadustat - placebo treatment difference

5. Secondary Outcome: Number (%) of Participants With Hb ≥10 g/dL Averaged Over Weeks 28 to 36 With Censoring for Rescue Therapy
Description: Hb values under the influence of a rescue therapy were censored by Cochran-Mantel-Haenszel Test for up to 6 weeks. Responder was defined as: Hb ≥10.0 g/dL, which was based on central laboratory values.
Time Frame: Weeks 28 to 36
Population: FAS Population consisted of all randomized/enrolled participants who received at least 1 dose of study drug and had baseline and at least 1 postdose Hb assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
Participants | 467 | 56
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 15.47, 95% CI 2-sided [10.79 to 22.189] — Roxadustat/placebo odds ratio

6. Secondary Outcome: Mean Change From Baseline in Low-Density Lipoprotein (LDL) Cholesterol Averaged Over Weeks 12 to 28
Description: Baseline LDL cholesterol was defined as the last LDL cholesterol value prior to the first dose of study drug.
Time Frame: Baseline (Day 1, Week 0), Weeks 12 to 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
mg/dL
  Baseline | 97.74 (39.09) | 96.39 (40.06)
  Change at Weeks 12 to 28: number analyzed (Participants) | 564 | 269
  Change at Weeks 12 to 28 | -18.48 (29.60) | 0.22 (29.37)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Treatment comparison was made using MMRM with baseline LDL cholesterol as a covariate, and treatment, visit, visit-by-treatment interaction, and the randomization stratification factors as fixed effects; Test type: Superiority; p < 0.0001, Mixed Models Analysis; MMRM Analysis; Least Square Mean Difference = -17.26, 95% CI 2-sided [-20.65 to -13.87], Standard Error of Mean 1.73 — Roxadustat- placebo treatment difference

7. Secondary Outcome: Rate of Change in eGFR From Baseline up to 12 Months (Linear Random Coefficient Model With Observed Data)
Description: Progression of chronic kidney disease was measured by rate of change in eGFR over time adjusted by baseline eGFR, with censoring for chronic dialysis or kidney transplant, using random slope and intercept model. Least Square Mean of change from baseline at 1 year was derived based on a random slopes and intercepts model using all available eGFR values (1 baseline and all post-treatment values up to end of treatment period + 7 days or start of dialysis) adjusted on treatment, baseline Hb, baseline eGFR, geographical region, cardiovascular events history at Baseline (yes vs. no), time (continuous value), the interaction terms of baseline eGFR by time, baseline Hb by time, and treatment by time as fixed effects, with random effects of intercept and linear slope of time. All assessments collected after the start of stable dialysis or kidney transplant were excluded from the analysis.
Time Frame: Baseline, Month 12
Population: FAS Population included all randomized/enrolled participants who received at least 1 dose of study drug and had baseline and at least 1 postdose Hb assessment.
Measure: Least Squares Mean (Standard Error); unit: ml/min/1.73 m^2
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
ml/min/1.73 m^2 | -2.89 (0.363) | -3.10 (0.388)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Test type: Superiority; p = 0.6924, ANCOVA; MI ANCOVA; Least Square Mean Difference = 0.21, 95% CI 2-sided [-0.827 to 1.245], Standard Error of Mean 0.528 — Roxadustat - placebo treatment difference

8. Secondary Outcome: Number of Participants Who Received Blood/RBC Transfusion in the First 52 Weeks of Treatment
Description: Participants with any use of blood/RBC transfusion were reported.
Time Frame: Baseline up to Week 52
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
Participants | 34 | 47
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Test type: Superiority; p < 0.0001, Cox Proportional hazards model — From a Cox Proportional hazards model adjusting for baseline Hb, baseline eGFR and other randomization stratification factors, except baseline Hb (≤8 g/dL versus >8 g/dL) and eGFR (<30 versus ≥30 mL/min/1.73 m^2); Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.165 to 0.406]

9. Secondary Outcome: Number (%) of Participants Who Received Rescue Therapy in the First 24 Weeks and in the First 52 Weeks of Treatment
Description: Rescue therapy included any use of RBC transfusion, ESA, or IV iron.
Time Frame: Baseline (Day 1, Week 0) up to Week 24 and up to Week 52
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
Participants
  24 Weeks | 29 | 61
  52 Weeks | 54 | 88
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; First 24 Weeks of Treatment; Test type: Superiority; p < 0.0001, Cox Proportional hazards model — From a Cox Proportional hazards model adjusting for baseline Hb, baseline eGFR and the randomization stratification factors, except baseline Hb (<=8 g/dL versus >8 g/dL) and eGFR (<30 versus >=30 mL/min/1.73m^2); Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0.108 to 0.267]
Statistical Analysis 2: Comparison: Roxadustat vs Placebo; First 52 Weeks of Treatment; Test type: Superiority; p < 0.0001, Cox Proportional hazards model — [p-value comment as in outcome 8, analysis 1]; Hazard Ratio (HR) = 0.19, 95% CI 2-sided [0.138 to 0.276]

10. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36) Version 2 Physical Functioning Subscore and Vitality Subscore at Weeks 12 to 28
Description: The SF-36 V2 consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems, role limitations due to emotional problems, general health perceptions, mental health, social function, and vitality. The physical functioning subscore and vitality subscore are reported. The scores ranged from 0 (worst) to 100 (Best). A higher score indicates a general improvement of life quality or well-being. Baseline score was defined as the last physical functioning value or vitality value, as applicable, prior to the first dose of study drug.
Time Frame: Baseline (Day 1, Week 0), Weeks 12 to 28
Population: FAS Population included all randomized/enrolled participants who received at least 1 dose of study drug and had baseline and at least 1 postdose Hb assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 605 | 302
scores on a scale
  Physical functioning subscore: Baseline | 41.16 (10.121) | 41.35 (10.070)
  Physical functioning subscore: Change at Weeks 12 to 28: number analyzed (Participants) | 558 | 266
  Physical functioning subscore: Change at Weeks 12 to 28 | 0.33 (7.302) | -0.27 (7.363)
  Vitality subscore: Baseline: number analyzed (Participants) | 604 | 302
  Vitality subscore: Baseline | 48.19 (10.146) | 47.62 (9.774)
  Vitality subscore: Change at Weeks 12 to 28: number analyzed (Participants) | 558 | 266
  Vitality subscore: Change at Weeks 12 to 28 | 1.90 (8.705) | 1.02 (8.334)

11. Secondary Outcome: Number (%) of Participants Who Experienced Exacerbation of Hypertension
Description: Exacerbation of hypertension was defined as an increase from baseline of ≥20 millimeter of mercury (mmHg) in systolic blood pressure (sBP) and sBP ≥170 mmHg or an increase from baseline of ≥15 mmHg in diastolic blood pressure (dBP) and dBP ≥110 mmHg.
Time Frame: Baseline up to Week 52
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
Participants | 140 | 48

12. Secondary Outcome: Mean Change From Baseline in Mean Arterial Pressure (MAP) Averaged Over Weeks 20 to 28
Description: Baseline MAP was defined as the last MAP value prior to the first dose of study drug.
Time Frame: Baseline, Weeks 20 to 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 608 | 305
mmHg
  Baseline | 92.16 (8.538) | 91.53 (8.077)
  Change at Weeks 20 to 28: number analyzed (Participants) | 546 | 243
  Change at Weeks 20 to 28 | 0.02 (8.648) | -0.12 (7.653)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1, Week 0) up to 28 days after the last dose of study drug (maximum treatment duration was 234.9 weeks for roxadustat and 208.1 weeks for placebo). Mortality presented is for the timeframe of Baseline (Day 1, Week 0) up to end of treatment (maximum treatment duration was 234.9 weeks for roxadustat and 208.1 weeks for placebo).
Description: The Safety Population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Roxadustat | Placebo
All-Cause Mortality (participants affected / at risk) | 38/611 | 11/305
Serious Adverse Events (participants affected / at risk) | 321/611 | 120/305
Other Adverse Events (participants affected / at risk) | 468/611 | 216/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Roxadustat (N=611) | Placebo (N=305)
Anemia (Blood and lymphatic system disorders) | 5 | 8
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 2
Acute myocardial infarction (Cardiac disorders) | 11 | 3
Angina pectoris (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 3 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 3 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 23 | 5
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 7 | 0
Myocardial ischaemia (Cardiac disorders) | 3 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 2 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 0
Choroidal neovascularisation (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal prolapse (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 0
Diabetic gastropathy (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal polyp (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 4 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 2 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 6 | 4
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 4 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 2 | 2
Catheter site haemorrhage (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Complication associated with device (General disorders) | 1 | 0
Device related thrombosis (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Medical device site irritation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 2
Pyrexia (General disorders) | 5 | 1
Terminal state (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic cyst ruptured (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Arteriovenous fistula site infection (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 3 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 1
Carbuncle (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 11 | 5
Cellulitis gangrenous (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 4 | 4
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 1
Kidney infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 6 | 0
Osteomyelitis acute (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 13 | 1
Pneumonia (Infections and infestations) | 29 | 12
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 2
Rectal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 8 | 0
Septic shock (Infections and infestations) | 5 | 0
Sinobronchitis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Ureteritis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 18 | 8
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 6 | 2
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 3 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Dialysis disequilibrium syndrome (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0
Femur fracture (Injury, poisoning and procedural complications) | 7 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Haemodilution (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 3 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 3 | 0
Troponin increased (Investigations) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 8 | 5
Gout (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 19 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 13 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 15 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 0
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Intracranial mass (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Post cardiac arrest syndrome (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Radicular pain (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 2
Tremor (Nervous system disorders) | 1 | 0
Uraemic encephalopathy (Nervous system disorders) | 3 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 41 | 6
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 13 | 5
Chronic kidney disease (Renal and urinary disorders) | 27 | 9
Diabetic end stage renal disease (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 2 | 0
End stage renal disease (Renal and urinary disorders) | 34 | 10
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal cyst ruptured (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 3 | 2
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/241 | 0/130 — This is a sex-specific adverse event that only affects male participants.
Ovarian cyst (Reproductive system and breast disorders) | 1/375 | 0/176 — This is a sex-specific adverse event that only affects female participants.
Prostatitis (Reproductive system and breast disorders) | 1/241 | 0/130 — This is a sex-specific adverse event that only affects male participants.
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Pleuroperitoneal communication (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypertensive crisis (Vascular disorders) | 4 | 1
Hypertensive emergency (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 2 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 2 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=611) | Placebo (N=305)
Anemia (Blood and lymphatic system disorders) | 12 | 39
Constipation (Gastrointestinal disorders) | 103 | 34
Nausea (Gastrointestinal disorders) | 85 | 29
Diarrhoea (Gastrointestinal disorders) | 77 | 31
Vomiting (Gastrointestinal disorders) | 52 | 20
Dyspepsia (Gastrointestinal disorders) | 38 | 12
Abdominal pain (Gastrointestinal disorders) | 32 | 13
Oedema peripheral (General disorders) | 89 | 28
Oedema (General disorders) | 48 | 9
Pyrexia (General disorders) | 36 | 8
Viral upper respiratory tract infection (Infections and infestations) | 97 | 40
Upper respiratory tract infection (Infections and infestations) | 78 | 48
Urinary tract infection (Infections and infestations) | 56 | 24
Bronchitis (Infections and infestations) | 33 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 98 | 38
Hypoglycemia (Metabolism and nutrition disorders) | 42 | 12
Decreased appetite (Metabolism and nutrition disorders) | 40 | 8
Hyperphosphatemia (Metabolism and nutrition disorders) | 40 | 10
Gout (Metabolism and nutrition disorders) | 32 | 20
Metabolic acidosis (Metabolism and nutrition disorders) | 26 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 54 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 23
Muscle spasms (Musculoskeletal and connective tissue disorders) | 41 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 39 | 14
Headache (Nervous system disorders) | 66 | 26
Dizziness (Nervous system disorders) | 57 | 32
Insomnia (Psychiatric disorders) | 62 | 9
End stage renal disease (Renal and urinary disorders) | 36 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 57 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 54 | 19
Hypertension (Vascular disorders) | 93 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen.

The investigator can only publish after the multisite consortium publishes (or tries to publish and fails).

FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT01750190/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT01750190/SAP_001.pdf